CLINICAL TRIAL: NCT04514991
Title: Healing After Endodontic Microsurgery Using Resorbable Collagen Based Bone Augmentation Material: A Randomized Controlled Clinical Trial
Brief Title: Bone Regenerative Techniques in Endodontic Microsurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 833538
Record Dates: First submitted 2020-07-31; First posted 2020-08-17 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Apical Periodontitis
Keywords: Persistent periapical pathology
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment (Experimental): Surgical sites (osteotomy) assigned to this group received endodontic microsurgery procedure+ Foundation (J. Morita USA).
  Interventions: Device: Foundation
- Control (No Intervention): Surgical sites (osteotomy) assigned to this group receives endodontic microsurgery procedure only.

INTERVENTIONS:
Device: Foundation — Collagen-based, bone filling augmentation material used to stimulate bone formation in extraction sockets or bone defects in the alveolar ridge.
  Arms: Treatment

SUMMARY:
The purpose of this randomized controlled clinical trial was to evaluate two dimensionally and 3-dimensionally the effect of resorbable collagen-based bone filling material on periapical healing following endodontic microsurgery (EMS) on endodontic lesions presenting four-wall defect.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult.
* Intact coronal restoration with no sign of leakage.
* Class B (small lesion) and C (large lesion) periapical lesions. (Kim and Kratchman 2006)

Exclusion Criteria:

* Patients with medical conditions and contraindications to surgery.
* Minors.
* Pregnancy.
* Teeth with signs of coronal leakage.
* Teeth with vertical root fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bekir Karabucak, DMD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- UPenn, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start date of recruitment: 09/03/2019 End date of recruitment: 12/15/2020
  Patients were consecutively enrolled until March 10th, 2020, after which all clinical and research activity was suspended due to the COVID-19 pandemic. The study was resumed in August 11th, 2020.
Units Other Than Participants: Osteotomy sites
Groups:
- Endodontic Microsurgery Only: Surgical sites assigned to this group receive Endodontic microsurgery procedure.
- Endodontic Microsurgery + Foundation: Surgical sites assigned to this group receive Endodontic microsurgery procedure+ Foundation (J. Morita USA).
  Foundation: Collagen-based, bone filling augmentation material used to stimulate bone formation in extraction sockets or bone defects in the alveolar ridge.
Period: Overall Study
Arm/Group | Endodontic Microsurgery Only | Endodontic Microsurgery + Foundation
Started | 41; 41 Osteotomy sites | 45; 45 Osteotomy sites
Completed | 30; 30 Osteotomy sites | 36; 36 Osteotomy sites
Not Completed | 11; 11 Osteotomy sites | 9; 9 Osteotomy sites

BASELINE CHARACTERISTICS:
Population: Randomization and analysis unit per periapical lesion . Some participants had multiple teeth with multiple lesions or multirooted teeth with separate lesions.
Units Other Than Participants: Lesions
Groups:
- Endodontic Microsurgery Only: Surgical sites assigned to this group received Endodontic microsurgery procedure.
- Foundation+ Endodontic Microsurgery: Surgical sites assigned to this group received Endodontic microsurgery procedure+ Foundation (J. Morita USA).
  Foundation: Collagen-based, bone filling augmentation material used to stimulate bone formation in extraction sockets or bone defects in the alveolar ridge.
- Total: Total of all reporting groups
Arm/Group | Endodontic Microsurgery Only | Foundation+ Endodontic Microsurgery | Total
Number analyzed (Participants) | 41 | 45 | 67
Number analyzed (Lesions) | 41 | 45 | 86
Age, Categorical [Count of Units; unit: Lesions] — Population: Randomization and analysis unit per periapical lesion . Some participants had multiple teeth with multiple lesions or multirooted teeth with separate lesions.
  Lesions
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 33 | 40 | 73
    >=65 years | 8 | 5 | 13
Sex: Female, Male [Count of Units; unit: Lesions]
  Female | 31 | 28 | 59
  Male | 10 | 17 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Arch [Count of Units; unit: Lesions]
  Maxilla | 26 | 29 | 55
  Mandible | 15 | 16 | 31
Tooth Type [Count of Units; unit: Lesions] — Population: Randomization and analysis unit per periapical lesion . Some participants had multiple teeth with multiple lesions or multirooted teeth with separate lesions.
  Lesions
    Anterior | 16 | 19 | 35
    Posterior | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: 2D Radiographic Healing at 12 Months Follow up (Overall Cases)
Description: Periapical healing was assessed by qualitatively evaluating bone regeneration through PA radiographs using well-established criteria. Molven's criteria categorize healing using periapical films into four categories: complete healing, incomplete healing, uncertain and unsatisfactory healing.
Time Frame: 12 months
Population: Analysis completed per osteotomy site.
Measure: Count of Units; unit: osteotomy site
Units Other Than Participants: osteotomy site
Groups:
- Control: Surgical sites assigned to this group received endodontic microsurgery procedure.
- Treatment: Surgical sites assigned to this group received endodontic microsurgery procedure+ Foundation (J. Morita USA).
  Foundation: Collagen-based, bone filling augmentation material used to stimulate bone formation in extraction sockets or bone defects in the alveolar ridge.
Arm/Group | Control | Treatment
Number analyzed (Participants) | 30 | 36
Number analyzed (osteotomy site) | 30 | 36
osteotomy site
  Complete healing | 24 | 29
  Incomplete healing | 1 | 1
  Uncertain healing | 3 | 3
  Unsatisfactory healing | 2 | 3

2. Primary Outcome: 3D Radiographic Healing at 12 Months Follow up (Overall Cases)
Description: Periapical healing was assessed by qualitatively evaluating bone regeneration through CBCT scans using Penn 3D criteria. Cases were classified into complete, limited, or unsatisfactory healing.
Time Frame: 12 months
Population: Analysis completed per osteotomy site.
Measure: Count of Units; unit: osteotomy sites
Units Other Than Participants: osteotomy sites
Groups:
- Foundation: Surgical sites assigned to this group receive endodontic microsurgery procedure+ Foundation (J. Morita USA).
  Foundation: Collagen-based, bone filling augmentation material used to stimulate bone formation in extraction sockets or bone defects in the alveolar ridge.
Arm/Group | Control | Foundation
Number analyzed (Participants) | 30 | 36
Number analyzed (osteotomy sites) | 30 | 36
osteotomy sites
  Complete | 11 | 22
  Limited | 14 | 10
  Unsatisfactory | 5 | 4

3. Primary Outcome: 2D Radiographic Healing at 12 Months Follow up (Asymptomatic Cases Only)
Description: as for outcome 1
Time Frame: 12 months
Population: Analysis per osteotomy. Excluded participants presenting with symptoms.
Measure: Count of Units; unit: osteotomy site
Units Other Than Participants: osteotomy site
Groups:
- Control: Surgical sites assigned to this group receive endodontic microsurgery procedure.
Arm/Group | Control | Foundation
Number analyzed (Participants) | 26 | 32
Number analyzed (osteotomy site) | 26 | 32
osteotomy site
  Complete | 23 | 28
  Incomplete | 1 | 1
  Uncertain | 1 | 2
  Unsatisfactory | 1 | 1

4. Primary Outcome: 3D Radiographic Healing at 12 Months Follow up (Asymptomatic Cases Only)
Description: as for outcome 2
Time Frame: 12 months
Population: Analysis per osteotomy site. Excluded participants with symptoms.
Measure: Count of Units; unit: osteotomy sites
Units Other Than Participants: osteotomy sites
Arm/Group | Control | Treatment
Number analyzed (Participants) | 26 | 32
Number analyzed (osteotomy sites) | 26 | 32
osteotomy sites
  Complete | 10 | 21
  Limited | 14 | 10
  Unsatisfactory | 2 | 1

5. Secondary Outcome: C Score (Overall Cases)
Description: Cortical plate healing using RAC/B index as evaluated on CBCT scans.
  Score 0: Cortical plate not re-established (Nonhealed). Score 1: Cortical plate is partially re-established (Partially healed). Score 2: Cortical plate is re-established (Completely healed).
Time Frame: 12 months
Population: Analysis per osteotomy site.
Measure: Count of Units; unit: osteotomy sites
Units Other Than Participants: osteotomy sites
Groups:
- Foundation: Surgical sites assigned to this group received endodontic microsurgery procedure+ Foundation (J. Morita USA).
  Foundation: Collagen-based, bone filling augmentation material used to stimulate bone formation in extraction sockets or bone defects in the alveolar ridge.
Arm/Group | Control | Foundation
Number analyzed (Participants) | 30 | 36
Number analyzed (osteotomy sites) | 30 | 36
osteotomy sites
  C-Score 2 | 13 | 23
  C-score 1 | 12 | 9
  C-score 0 | 5 | 4

6. Secondary Outcome: C Score (Asymptomatic Cases Only)
Description: as for outcome 5
Time Frame: 12 months
Population: Analysis per osteotomy site. Excluded participants with symptoms.
Measure: Count of Units; unit: osteotomy sites
Units Other Than Participants: osteotomy sites
Arm/Group | Control | Foundation
Number analyzed (Participants) | 26 | 32
Number analyzed (osteotomy sites) | 26 | 32
osteotomy sites
  C-score 2 | 12 | 22
  C-score 1 | 12 | 9
  C-score 0 | 2 | 1

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Groups:
- Endodontic Microsurgery: Surgical sites assigned to this group received endodontic microsurgery procedure.
- Endodontic Microsurgery + Foundation: Surgical sites assigned to this group received endodontic microsurgery procedure+ Foundation (J. Morita USA).
  Foundation: Collagen-based, bone filling augmentation material used to stimulate bone formation in extraction sockets or bone defects in the alveolar ridge.
Arm/Group | Endodontic Microsurgery | Endodontic Microsurgery + Foundation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT04514991/Prot_SAP_001.pdf